CLINICAL TRIAL: NCT07395271
Title: Comparing Doses of Intrathecal Dexmedetomidine Along With Bupivacaine for Cesarean Section: A Double-Blind Randomized Clinical Trial
Brief Title: Comparing Doses of Intrathecal Dexmedetomidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bahria International Hospital (Unknown)
Responsible Party: Principal Investigator, Azher Munir, Principal Investigator, Postgraduate Resident, Bahria International Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2021-6907
Record Dates: First submitted 2026-01-23; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Dexmedetomidine
Keywords: Dexmedetomidine; spinal anesthesia; cesarean section; bupivacaine; sensory block; motor block
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Dexmedetomidine 5 mcg
  Interventions: Drug: Dexmedetomidine 5 mcg
- Group B (Active Comparator): Dexmedetomidine 10 mcg
  Interventions: Drug: Dexmedetomidine 10 mcg

INTERVENTIONS:
Drug: Dexmedetomidine 5 mcg — 12.5 mg (2.5 mL) of 0.5% hyperbaric bupivacaine + 5 µg dexmedetomidine
  Other Names: Dexmedetomidine 5mcg
  Arms: Group A
Drug: Dexmedetomidine 10 mcg — 12.5 mg (2.5 mL) of 0.5% hyperbaric bupivacaine + 10 µg dexmedetomidine
  Other Names: Dexmedetomidine 10mcg
  Arms: Group B

SUMMARY:
To compare the duration of sensory and motor blockade produced by two different intrathecal doses of dexmedetomidine (5 µg and 10 µg) when added to hyperbaric bupivacaine in patients undergoing elective cesarean section

DETAILED DESCRIPTION:
Cesarean section remains one of the most commonly performed surgical procedures worldwide, serving as a critical intervention to reduce maternal and neonatal morbidity when vaginal delivery poses increased risks. Global cesarean delivery rates have risen steadily, from approximately 7% in 1990 to around 21% in recent years, with projections indicating that by 2030, nearly one in three births may occur via cesarean section .This trend is particularly pronounced in regions like Latin America and the Caribbean (over 40%) and varies significantly by socioeconomic factors, healthcare access, and clinical indications . In Pakistan and similar settings, rates continue to increase, underscoring the need for optimized anesthetic techniques that prioritize maternal safety, fetal well-being, rapid recovery, and effective postoperative pain control.

Regional anesthesia, specifically spinal anesthesia, is the preferred method for elective cesarean sections due to its rapid onset, avoidance of airway complications associated with general anesthesia, minimal placental transfer of drugs, and enhanced maternal satisfaction. Hyperbaric bupivacaine is the most widely used local anesthetic for this purpose, providing reliable sensory and motor blockade. However, when used alone, bupivacaine offers relatively short-duration postoperative analgesia, which can delay ambulation, hinder early mother-infant bonding, and increase the need for systemic analgesics6. To address these limitations, various intrathecal adjuvants have been investigated to enhance block quality, prolong analgesia, and improve overall outcomes.

Dexmedetomidine, a highly selective α2-adrenergic agonist, exhibits sedative, anxiolytic, and analgesic properties without significant respiratory depression. When administered intrathecally, it inhibits nociceptive transmission through presynaptic C-fibers and postsynaptic dorsal horn neurons, resulting in prolonged sensory and motor blockade compared to bupivacaine alone8,9 . Multiple recent studies and meta-analyses have confirmed its efficacy as an adjuvant in obstetric spinal anesthesia, demonstrating extended analgesia duration, reduced shivering, and fewer side effects (e.g., pruritus, nausea) than opioids like fentanyl . However, the optimal intrathecal dose remains controversial: lower doses (e.g., 3-5 µg) may offer a favorable benefit-risk profile with minimal hemodynamic impact, while higher doses (e.g., 10 µg) provide greater prolongation but raise concerns about potential bradycardia or hypotension in parturient.

This prospective, double-blind, randomized clinical trial compares the effects of two commonly used doses of intrathecal dexmedetomidine-5 µg and 10 µg-when added to a standard dose of hyperbaric bupivacaine (12.5 mg) for elective cesarean section. The primary aim is to determine which dose yields superior prolongation of sensory and motor blockade while maintaining maternal hemodynamic stability and safety.

ELIGIBILITY:
Inclusion Criteria:

* Parturients aged 20-40 years
* ASA physical status II
* Scheduled for elective cesarean section
* Ability to provide informed written consent

Exclusion Criteria:

* ASA physical status III or higher
* Emergency cesarean section
* Previous labor analgesia
* History of cardiovascular, neurological, or systemic disease
* Contraindications to spinal anesthesia
* Surgery duration exceeding 60 minutes

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Duration of sensory blockade | 6 hrs
  Visual Analouge Scale (0 to 10)
Duration of motor blockade | 6 hrs
  Bromage Scale (1 to 5)

SECONDARY OUTCOMES:
Hemodynamic parameters | Till end of surgery
  Heart rate per minute
Hemodynamic parameters | Till end of surgery
  Mean arterial pressure in millimeters of mercury

CONTACTS AND LOCATIONS:
Overall Officials: azher munir, mbbs, Principal Investigator — Bahria International Hospital
Locations (1):
- Bahria International Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mowar A, Singh V, Pahade A, Karki G. Effect of three different doses of intrathecal dexmedetomidine on subarachnoid block: a prospective randomized double-blind trial. Anaesth. pain intensive care 2021;26(1):8-13; DOI:10.35975/apic.v26i1.1759